CLINICAL TRIAL: NCT03695991
Title: Effect of Per-cutaneous Nephrosotomy Drainage on Radioisotope Imaging of Hydronephrotic Kidneys
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Atef Ali, Principal investigator, Assiut University
Other Study IDs: PCNHK
Record Dates: First submitted 2018-10-03; First posted 2018-10-04 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Hydronephrosis
MeSH Terms: conditions — Hydronephrosis | interventions — Nephrostomy, Percutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients will be recruited from out-patient clinics and in-patient sectors of Assiut Urology and Nephrology hospital
  Interventions: Procedure: percutaneous nephrostomy

INTERVENTIONS:
Procedure: percutaneous nephrostomy — The percutaneous nephrostomy will be done under sonographic or fluoroscopic guidance. Establishment of intravenous access and antibiotics will be performed half an hour prior to procedure particularly in patients presenting with urinary tract infection. The procedure will be done under local anesthesia but general anesthesia may be used for uncooperative patients. percutaneous nephrostomy will be performed in the prone position, however, in case of relative contraindication to prone position

SUMMARY:
Hydronephrosis describes a condition of urine-filled dilation of the collecting system. Normally, urine flows through the urinary tract with minimal or low pressure. If the build-up of excess fluid in the urinary collecting system continues, there will be an increase in pressure and atrophy of renal cortex. If hydronephrosis is left untreated for a long time, renal damage with permanent loss of function occurs

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients for whom a percutaneous nephrostomy is indicated provided that the hydronephrosis is advanced ( parenchymal thickness not more than 5 mm ) 2) Patients for whom a nephrectomy is planned for a seemingly poorly functioning kidney along with either

Exclusion Criteria:

1. Target kidney is the only functioning or better functioning kidney or otherwise substantially contributing to the total renal function, so nephrectomy is not likely.
2. Emergency cases where the general condition of the patient cannot withstand the logistics of undergoing a radioisotope study eg
3. Malignancy in the target kidney
4. Patients unlikely to undergo a nephrectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited from out-patient clinics and in-patient sectors of Assiut Urology and Nephrology hospital
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The rate of increase in glomerular filtration rate after intervention | 3 weeks
  the radioisotope measurement of glomerular filtration rate will be done before and after insertion of percutaneous nephrostomy tube